CLINICAL TRIAL: NCT06262685
Title: A Multicenter, Controlled, Randomized, Single-blind Phase IV Trial Assesses Efficacy, Safety, and Cost of Pre-emptive Genotyping in a Cardiovascular Risk Population Eligible for High/Moderate-intensity Statins
Brief Title: Efficacy, Safety and Cost-efficacy of a Pre-emptive Genotyping Strategy in Patients Receiving Statins
Acronym: PREVESTATGx
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-509418-12-00
Record Dates: First submitted 2024-01-09; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Dyslipidemias; Statin Adverse Reaction; Pharmacogenic Myopathy
Keywords: Statin; Statin Associated Muscle Symptoms; Cardiovascular disease; Cost-effectiveness; Phase IV Clinical Trial; Pharmacogenetic
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias; Malignant fever | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Phase IV, multicentre, controlled, randomized, parallel and single-blind adaptive clinical trial nested within the iPHARMGx master protocol study
Who Masked: Participant
Masking Description: Subjects will remain blinded to arm assigned because pharmacogenetic phenotype and statin/dose-guidance will only be exclusively accesible to the attending physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients in this Experimental Group will receive any of the statins authorized in Spain for lipid-lowering, both for primary and secondary prevention. Subjects in the Experimental Group will be administered the specific type and dosage of statins recommended by the Clinical Pharmacogenetics Consortium's genotype guidelines, utilizing the patient's pharmacogenetic information and characteristics
  Interventions: Other: Preemptive pharmacogenetic atorvastatin dose based on CPIC guidelines; Other: Preemptive pharmacogenetic simvastatin dose based on CPIC guidelines; Other: Preemptive pharmacogenetic pitavastatin dose based on CPIC guidelines; Other: Preemptive pharmacogenetic rosuvastatin dose based on CPIC guidelines; Other: Preemptive pharmacogenetic pravastatin dose based on CPIC guidelines; Other: Preemptive pharmacogenetic lovastatin dose based on CPIC guidelines; Other: Preemptive pharmacogenetic fluvastatin dose based on CPIC guidelines
- Control Group (Active Comparator): Patients in this Control Group will receive any of the authorized statins in Spain for lipid-lowering, whether for primary or secondary prevention. They will be administered statins according to clinical practice and the drug's product labeling, without exceeding the already authorized dosages
  Interventions: Other: Standard of Care (SoC) dosing of atorvastatin; Other: Standard of Care (SoC) dosing of simvastatin; Other: Standard of Care (SoC) dosing of pitavastatin; Other: Standard of Care (SoC) dosing of rosuvastatin; Other: Standard of Care (SoC) dosing of prasavastatin; Other: Standard of Care (SoC) dosing of lovastatin; Other: Standard of Care (SoC) dosing of fluvastatin

INTERVENTIONS:
Other: Preemptive pharmacogenetic atorvastatin dose based on CPIC guidelines — Atorvastatin at the dosage reccomended by the 2022 "Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for SLCO1B1, ABCG2, and CYP2C9 genotypes and considerations for Statin-Associated Musculoskeletal Symptoms" based on the subjects pharmacogenetic phenotype. A comprehensive description of said doses are can be accessed at: https://cpicpgx.org/guidelines/cpic-guideline-for-statins/
  Arms: Experimental Group
Other: Preemptive pharmacogenetic simvastatin dose based on CPIC guidelines — Simvastatin at the dosage reccomended by the 2022 "Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for SLCO1B1, ABCG2, and CYP2C9 genotypes and considerations for Statin-Associated Musculoskeletal Symptoms" based on the subjects pharmacogenetic phenotype. A comprehensive description of said doses are can be accessed at: https://cpicpgx.org/guidelines/cpic-guideline-for-statins/
  Arms: Experimental Group
Other: Preemptive pharmacogenetic pitavastatin dose based on CPIC guidelines — Pitavastatin at the dosage reccomended by the 2022 "Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for SLCO1B1, ABCG2, and CYP2C9 genotypes and considerations for Statin-Associated Musculoskeletal Symptoms" based on the subjects pharmacogenetic phenotype. A comprehensive description of said doses are can be accessed at: https://cpicpgx.org/guidelines/cpic-guideline-for-statins/
  Arms: Experimental Group
Other: Preemptive pharmacogenetic rosuvastatin dose based on CPIC guidelines — Rosuvastatin at the dosage reccomended by the 2022 "Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for SLCO1B1, ABCG2, and CYP2C9 genotypes and considerations for Statin-Associated Musculoskeletal Symptoms" based on the subjects pharmacogenetic phenotype. A comprehensive description of said doses are can be accessed at: https://cpicpgx.org/guidelines/cpic-guideline-for-statins/
  Arms: Experimental Group
Other: Preemptive pharmacogenetic pravastatin dose based on CPIC guidelines — Pravastatin at the dosage reccomended by the 2022 "Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for SLCO1B1, ABCG2, and CYP2C9 genotypes and considerations for Statin-Associated Musculoskeletal Symptoms" based on the subjects pharmacogenetic phenotype. A comprehensive description of said doses are can be accessed at: https://cpicpgx.org/guidelines/cpic-guideline-for-statins/
  Arms: Experimental Group
Other: Preemptive pharmacogenetic lovastatin dose based on CPIC guidelines — Lovastatin at the dosage reccomended by the 2022 "Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for SLCO1B1, ABCG2, and CYP2C9 genotypes and considerations for Statin-Associated Musculoskeletal Symptoms" based on the subjects pharmacogenetic phenotype. A comprehensive description of said doses are can be accessed at: https://cpicpgx.org/guidelines/cpic-guideline-for-statins/
  Arms: Experimental Group
Other: Preemptive pharmacogenetic fluvastatin dose based on CPIC guidelines — Fluvastatin at the dosage reccomended by the 2022 "Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for SLCO1B1, ABCG2, and CYP2C9 genotypes and considerations for Statin-Associated Musculoskeletal Symptoms" based on the subjects pharmacogenetic phenotype. A comprehensive description of said doses are can be accessed at: https://cpicpgx.org/guidelines/cpic-guideline-for-statins/
  Arms: Experimental Group
Other: Standard of Care (SoC) dosing of atorvastatin — Subject allocated to this arm will receive the atorvastatin according to clinical practice and the drug's product labelling, and never exceeding the already authorized dosages. These subject will not receive a personalised dosed/prescription based on their pharmacogenetic phenotype
  Arms: Control Group
Other: Standard of Care (SoC) dosing of simvastatin — Subject allocated to this arm will receive the simvastatin according to clinical practice and the drug's product labelling, and never exceeding the already authorized dosages. These subject will not receive a personalised dosed/prescription based on their pharmacogenetic phenotype
  Arms: Control Group
Other: Standard of Care (SoC) dosing of pitavastatin — Subject allocated to this arm will receive the pitavastatin according to clinical practice and the drug's product labelling, and never exceeding the already authorized dosages. These subject will not receive a personalised dosed/prescription based on their pharmacogenetic phenotype
  Arms: Control Group
Other: Standard of Care (SoC) dosing of rosuvastatin — Subject allocated to this arm will receive the rosuvastatin according to clinical practice and the drug's product labelling, and never exceeding the already authorized dosages. These subject will not receive a personalised dosed/prescription based on their pharmacogenetic phenotype
  Arms: Control Group
Other: Standard of Care (SoC) dosing of prasavastatin — Subject allocated to this arm will receive the prasavastatin according to clinical practice and the drug's product labelling, and never exceeding the already authorized dosages. These subject will not receive a personalised dosed/prescription based on their pharmacogenetic phenotype.
  Arms: Control Group
Other: Standard of Care (SoC) dosing of lovastatin — Subject allocated to this arm will receive the lovastatin according to clinical practice and the drug's product labelling, and never exceeding the already authorized dosages. These subject will not receive a personalised dosed/prescription based on their pharmacogenetic phenotype.
  Arms: Control Group
Other: Standard of Care (SoC) dosing of fluvastatin — Subject allocated to this arm will receive the fluvastatin according to clinical practice and the drug's product labelling, and never exceeding the already authorized dosages. These subject will not receive a personalised dosed/prescription based on their pharmacogenetic phenotype.
  Arms: Control Group

SUMMARY:
This is a Phase IV multicentre adaptive single-blinded randomized clinical trial if preemptively genotyping populations at risk of cardiovascular disease susceptible of receiving high or moderate doses of statin therapy is efficacious, cost-efficacious, and feasible within the Spanish National Health System when compared to the current standard of care. This trial is nested within the iPHARMGx master protocol

DETAILED DESCRIPTION:
This is a nation-wide, multicentre, randomised, controlled, and adaptive phase IV clinical trial that aims to assess the efficacy and cost-efficacy of pre-emptive pharmacogenetic testing strategies, including those impacted by genetic variants associated with adverse drug reactions (ADRs) or limited efficacy. Populations at high-risk of developing clinically relevant outcomes will be enrolled in nested trials within this master protocol. The clinical trials will evaluate the efficacy and cost-efficacy of pre-emptive genotyping by defining a drug-gene-endpoint triad. Study subjects will be pre-emptively genotyped and, if found to have an actionable gene variant, randomly allocated to either a test group where guideline-based treatment modifications will be initiated or a control group that will be managed according to healthcare provider standard of care (SoC). Subsequently, subjects will be prospectively followed at prespecified timepoints. Detailed information on drug-gene-endpoint triads, allocation schemes, and follow-up visits will be provided in each of the subprotocols. A Data Monitoring Committee (DMC), composed of physician experts, will be appointed for each nested trial to review the data on an ongoing basis, ensuring the safety of participants and scientific validity of the study.

ELIGIBILITY:
Inclusion Criteria:

Each potential participant must satisfy all of the following criteria to be enrolled in the study:

1. Ability of the participant to understand the purpose and risks of the study, to provide informed consent, and to authorize the use of confidential health information in accordance with national and local privacy regulations.
2. Subject has voluntarily signed the ICF.
3. Subject must be ≥ 18 years old at the time of signing ICF.
4. Subject is able and willing to take part and be followed-up for the majority of the study duration.
5. Participants are susceptible to be prescribed any of the following:

   1. Atorvastatin ≥40 mg/day p.o.
   2. Simvastatin ≥20mg/day p.o.
   3. Pitavastatin≥2mg/day p.o.
   4. Rosuvastatin ≥40mg/day p.o.
   5. Pravastatin ≥40mg/day p.o.
   6. Lovastatin ≥40mg/day p.o.
   7. Fluvastatin ≥80 mg/day p.o.
6. Subjects must be naïve to any genotyping test of the following genes: SCLO1B1, ABCG2, CYP2C9, CYP3A4, CYP3A5 and HMGCR.
7. Subjects must be willing to comply and adhere to any treatment plan modifications established and to the procedures specified in this protocol.
8. Women of childbearing potential must commit not to become pregnant. Subjects must be willing to use highly effective contraceptive methods or have practiced sexual abstinence during the study.

Exclusion Criteria:

Any potential participant who meets any of the following criteria will be excluded from participating in the study:

1. Subject is currently taking ubiquinone (Q10) supplements.
2. Known personal or family history of statin-associated autoimmune myopathy or HMG-CoA reductase disorder.
3. Pregnant or breastfeeding women
4. Subject has a personal history or analytical evidence of one of the following disorders:

   1. Any contraindications to statin administration as revealed in the summary of product characteristics (SmPCs) for statins.
   2. Prior SAMS if subject is not statin-naïve.
5. Any condition or situation deemed by the investigator precluding or interfering with the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-03-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically relevant statin-associated musculoskeletal events | 9-months
  As defined by the a composite endpoint:
  Patients with a clinically relevant statin-associated musculoskeletal symptom defined as a combination of a SAMS-CI (Statin Associated Muscular Symptoms Clinical Index) score ≥7 points and a NPRS (Numerical Pain Rating Scale) score ≥3) in the 9-month follow-up period
  Serum creatin phosphokinase (CPK) [UI/L] greater than three times the upper limit of normality prespecified by each centre's laboratory, in relation to the statin.

SECONDARY OUTCOMES:
Low density lipoprotein cholesterol (LDLc) serum concentration baseline reduction rate | 9-months
  Percentage of Baseline LDLc serum concentration reduction rate when compared to LDLc serum concentration values at 9 months.
Baseline change in statin therapy prescription | 9-months
  Percentage of patients that require either a statin dose modification/withdrawal or additional lipid-lowering therapy after 9 months in order to meet LDLc goals.
Cost of a statin preemptive pharmacogenetic prescription scheme | Though study completion, on average 18 months
  To quantify economic burden a cost-benefit analysis defined as the difference [in monetary units, euros] between the costs of the intervention [pharmacogenetic analysis] and all its surrounding procedures [personnel, geneticist report, clinical pharmacologist report] combined with the costs derived from the events [blood sample analysis, hospital admission, follow-up visits, lipid-lowering therapy modification] in the intervention arm when compared to the costs derived from the events in the control arm alone
  Monetary units requiered to prevent a event will be calculated through an incremental cost effectiveness ratio (ICER) between intervention and control arm .

OTHER OUTCOMES:
Novel prognostic and predictive genetic biomarkers of statin-related adverse events and efficacy identification | Though study completion, on average 18 months
  All participants DNA sample will be susceptible of deep sequencing analysis at CNIO (National Centre of Oncological Investigations) to assess novel prognostic and predictive biomarkers for statin induced muscle symptoms such as fibroblast growth factor 21 (FGF21), MicroRNA-499 or IL-6.
Death from cardiovascular causes, nonfatal myocardial infarction or hospitalization for unstable angina or resuscitated cardiac arrest | 9-months
  Combined incidence of participants who experience a 4-component exploratory endpoint consisting of:
  Cardiovascular death Nonfatal myocardial infarction (MI) Resuscitated cardiac arrest Hospitalization for unstable angina
Difference in percentage in the eight-item Morisky Medication Adherence Scale (MMAS-8) questionnaire score between intervention and control arm | 9-months
  A score <6 indicates low adherence A score of 6-8 indicates medium adherence A score >8 indicates high adherence
SAMS intensity reduction of a statin preemptive pharmacogenetic prescription scheme | 9-months
  Difference in Numeric Pain Rating Scale (NPRS) score between intervention and control arm.
  Categories will be as follow: 0-3 no pain; 3-5 moderate pain; 5-7 intense pain; 7-9 very intense pain; 9-10 extreme pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
A copy of the database of data collected during the clinical trial will be attached as an appendix to the publication resulting from this clinical trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available at the same time as the results will be published, and will be kept available to everyone without any time limit.
Access Criteria: Data will be available indefinitely on the publisher's website, as long as it is kept by the Publisher, for anyone who wishes to access the data, for non-commercial purposes

REFERENCES:
- [Derived] Stewart S, Seco-Meseguer E, Diago-Sempere E, Marin-Candon A, Carmona M, Estebanez M, Lopez-Fernandez LA, Imaz-Iglesia I, Del Mar Garcia Saiz M, Laserna-Mendieta EJ, Peiro AM, Farre M, Rodriguez-Jimenez C, Saiz-Rodriguez M, Sanabria-Cabrera J, Rosas-Alonso R, Abad-Santos F, Pedrosa L, Carcas AJ, Garcia Garcia I, Borobia AM; iPHARMGx study group. Phase IV adaptive randomised clinical trials evaluating efficacy and cost-efficacy of pre-emptive pharmacogenetic genotyping strategies in the Spanish National Health System: iPHARMGx Master Protocol and PREVESTATGx nested clinical trial. BMJ Open. 2024 Nov 7;14(11):e089823. doi: 10.1136/bmjopen-2024-089823. PMID 39510769